CLINICAL TRIAL: NCT07301398
Title: Construction and Preliminary Validation of a Community Health Education Program for Patients With Interstitial Lung Disease Based on Mobile Healthcare
Brief Title: Development & Preliminary Validation of a Community Health Education Program
Status: Not yet recruiting | Type: Observational
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2025-126
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Non-neoplastic and Non-infectious Diseases
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Intervention Measures for the Control Group: Patients in the control group received interventions through routine health education, telephone follow-up, and questionnaire surveys during follow-up visits. Health education covered disease-related knowledge, medication guidance, rehabilitation guidance, dietary guidance, and psychological guidance. After discharge, patients were followed up once a month via telephone or home visit, and questionnaire data were collected during their follow-up consultations.
- Experimental Group: Intervention Measures for the Experimental Group: On the basis of routine health education, the experimental group additionally received guidance on the use of the mini-program. Patients were instructed to proficiently use the mini-program's functions, including accessing health education information, interacting with medical staff, and understanding the precautions for questionnaire completion, and were advised to fill out the questionnaire monthly. Doctors and nurses were guided to master the mini-program to irregularly push health education-related knowledge to patients, and medical staff were instructed on the effective collection of questionnaire data and data statistics.
  Interventions: Behavioral: The use and guidance of the mini-program

INTERVENTIONS:
Behavioral: The use and guidance of the mini-program — Interventions were conducted through routine health education, telephone follow-ups, and questionnaire surveys during reconsultations. Health education covered disease knowledge, medication guidance, rehabilitation guidance, dietary guidance, and psychological guidance. After discharge, patients were followed up by telephone or home visit once a month, and questionnaire data were collected during their reconsultations. The use of a mini-program was added with corresponding guidance: patients were instructed to proficiently use the mini-program's functions for accessing health education information, interacting with medical staff, and noting key points for questionnaire completion, and were advised to fill out the questionnaire monthly. Doctors and nurses were guided to skillfully use the mini-program to push health education-related knowledge to patients at irregular intervals, and medical staff were trained on the effective collection of questionnaire data and data statistics.
  Groups: Experimental Group

SUMMARY:
This study analyzes the needs of patients regarding the content and form of home-based health education through interviews, and constructs a health education program tailored to these needs. A practical WeChat mini-program is developed to enable patients with interstitial lung disease to promptly access comprehensive health education information, consult about follow-up visits, and check test reports during their home care period, ultimately aiming to improve patients' quality of life and reduce medical consumption.

DETAILED DESCRIPTION:
Interstitial Lung Disease (ILD) refers to a group of non-neoplastic and non-infectious diseases primarily affecting the alveolar walls, including lesions in the perialveolar tissues and adjacent supporting structures. It is characterized by progressive dyspnea, deteriorating lung function, and poor prognosis. In recent years, with the deterioration of air quality, the continuous advancement of diagnosis and treatment technologies, and physicians' deepened understanding of ILD, the diagnosis rate of ILD has been increasing year by year. As the detection rate rises, growing attention is paid to the survival and treatment of ILD patients.

ILD patients often experience labored and rapid breathing, which limits their ability to perform daily activities. Low levels of physical function and vitality, coupled with severe dyspnea and fatigue, lead to a poor quality of life for these patients. Currently, clinical treatments can only control disease progression to a certain extent. Enhancing ILD patients' knowledge of their condition, encouraging active participation of patients and their families in nursing care, and improving patients' ability to monitor and manage their own health can effectively reduce the risk of infections, ensure the clinical efficacy of implemented treatment plans, and further alleviate patients' clinical symptoms.

With societal progress and advances in medical technology, telemedicine has gradually been applied in clinical practice. Telemedicine interventions have proven beneficial for the home-based management and control of chronic diseases such as hypertension and diabetes. Therefore, integrating telemedicine with existing medical and nursing approaches for the home-based health guidance of ILD patients constitutes an innovative research with significant scientific value.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with interstitial lung disease; Aged 18 years or older; Patients who have given informed consent to participate in this study; Proficient in Chinese with no comprehension barriers; Capable of independently using internet-enabled mobile devices.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Complicated with other life-threatening diseases; Consciousness disturbance or mental illness; Currently participating in other clinical trials that may affect this study.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Improve patients' quality of life and reduce medical consumption | One year after the start of recruitment
  Guide doctors and nurses to proficiently use the mini-program to push health education-related knowledge to patients at irregular intervals, and instruct medical staff on the effective collection of questionnaire data and data statistics.

IPD SHARING:
Plan to Share IPD: No